CLINICAL TRIAL: NCT05826743
Title: Safety and Effectiveness Evaluations of the COLO-BT™ (Colorectal Balloon Tube) as an Alternative Treatment to the Temporary Ileostomy Following Proctectomy
Brief Title: Safety and Effectiveness Evaluation of the COLO-BT as an Alternative Treatment to the Ileostomy
Acronym: COLO-BT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JSR Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSR CB
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Surgery; Colorectal Cancer; Rectal/Anal; Ileostomy - Stoma; Anastomotic Leakage
Keywords: Colorectal Surgery; Colorectal Cancer; Stoma; ileostomy; Anastomotic leakage
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- COLO BT™ (Experimental): Patients receive COLO BT™ during colorectal surgery.
  Interventions: Device: COLO BT™
- Standard of Care (Active Comparator): Patients receive the standard of care, a protective stoma, during colorectal surgery.
  Interventions: Other: Stoma Creation

INTERVENTIONS:
Device: COLO BT™ — A removable, temporary intraluminal bypass device designed to safely postpone the creation of a protective stoma after surgery for only patients who need it (do not have a healed anastomosis)
  Other Names: COLO BT
  Arms: COLO BT™
Other: Stoma Creation — Protective ileostomy
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate the Colorectal Balloon Tube (hereinafter referred to as COLO-BT™) device, a single use, temporary intraluminal bypass device, intended to reduce contact of fecal content with an anastomotic site, following colorectal surgery (open or laparoscopic)

DETAILED DESCRIPTION:
A primary diverting stoma is widely used by surgeons in order to bypass low rectal anastomosis and reduce morbidity associated with anastomotic leaks. Typically, a stoma is created for all high-risk patients which mean that many patients are exposed to potentially serious complications associated with the stoma itself without any clinical benefit.

COLO BT™ is a local, temporary bypass device that provides protection of the anastomosis and safely postpones stoma. COLO BT™ is designed to avoid stoma creation in all patients except those patients whose anastomoses have not healed after surgery, allowing the others to return to normal activity more quickly and safely.

ELIGIBILITY:
Inclusion Criteria:

The patient must meet all study Inclusion Criteria as outlined below:

* Adult males or females, 19-80 years of age, with signed informed consent

  * Subject whose anastomosis is expected to be located above 4cm from the anus, and at or below 15cm from the anus. (4cm < inclusion target ≤ 15cm from the anus).

    ③ Patient must meet all other inclusion criteria to be eligible. While not required, if one or more of the following six risk factors for postoperative anastomotic leakage[6,7,8] is true, the patient will be considered a high-risk subject:

    - Male

    - Those with a body mass index of 30 or higher

    - Current smoker

    - Those who are on medication for diabetes

    - Those with clinical stage III or higher malignant tumors

    - Those who received chemo/radiation therapy before surgery

    ④ Those who are willing and able to participate in this clinical study, provide Informed Consent, and are willing to comply with the study procedures and follow up evaluations

    ⑤ Those who have willingness to undertake blood transfusion if required.

Exclusion Criteria:

Patients meeting any of the following Exclusion Criteria will not be eligible to participate in the study:

1. Women who are pregnant or breastfeeding
2. Those who receive emergency surgery
3. A person who is expected to need intensive medical care after the surgery due to a serious medical condition, with one or more of the following seven factors being true:

   * Patients with abnormal bone marrow function (those with hemoglobin less than 7g/dl, leukocyte count less than 4000/mm3, or platelet count less than 100,000/mm3 even after preoperative corrections)
   * Patients with severe liver damage or cirrhosis (those whose AST/ALT levels are more than three times the normal range or those diagnosed with cirrhosis)
   * Those with abnormal renal function (those who are on hemodialysis or who have a blood creatinine level of 2.0mg/dl or more before the surgery)
   * Those who have undergone cardiac or cerebrovascular stent procedure within the last 6 months
   * Those who have been diagnosed with pulmonary tuberculosis within the last 6 months or are undergoing drug treatment for pulmonary tuberculosis
   * Those who continuously administer steroids of 20mg/day or more within 30 days before the surgery
   * Patients with ASA (American Society of Anesthesiologists) score of 3 are evaluated by the investigator who determines whether or not patients with ASA score of 3 should be enrolled from the patient safety standpoint. Patients with ASA score higher than 3 are excluded from this study.
   * Patients who are required to undergo re-intervention to treat the anastomosis following intraoperative positive air leak test (However, patients who underwent complete reconstruction of the anastomosis in the presence of a positive air test, which therefore has made their risk of leak similar to those patients with a negative air leak test.)
   * Patients who are immune suppressed
   * Patients with severe diverticulosis
   * Patients with other colonic wall abnormalities in the likely area of the Outer Balloon and BT BAND application who may be at increased risk for device perforation or migration.
4. A person who has difficulty in mobility or is unable to communicate in general due to a psychiatric/neurologic disorder falling under one or more of the following:

   * Those diagnosed with dementia or Alzheimer's disease.
   * Those who have been diagnosed with schizophrenia or depression or are taking drugs due to this.
   * A person who has been diagnosed with disability due to intellectual disability.
5. Patients with intestinal perforation, abscess in the pelvis, or severe inflammation in the pelvis.
6. Those who have a history of undergoing major surgeries (major bowel resection/major gastrectomy, major hepatectomy) through laparotomy and are likely to have serious adhesions that may affect this surgery.
7. A patient who underwent a preoperative chemotherapy, but the anastomosis is expected to be located very close to the anus or in the anal canal, thus with a very high risk for complications of the anastomosis, or a patient whom the bowel function is expected to decrease significantly in the future.
8. Patients who had pre-operative radiotherapy should be excluded.
9. Patients with inflammatory bowel diseases such as ulcerative colitis, Crohn's disease, intestinal tuberculosis, or autoimmune diseases such as Bechet's disease.
10. Those who do not consent in writing to the study.
11. Experienced blood loss (>750 cc) within 6 weeks before randomization.
12. Transfusion during surgery.
13. Any new sign of ischemia within 6 weeks before randomization.
14. Diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, intraabdominal infection, ischemic bowel all due to carcinomatosis within 6 weeks before randomization.
15. Known hypersensitivity or allergy to any of the components required for the procedure.
16. Exclusion criteria not specified above, but the patient is determined to be unsuitable for participation in this clinical study at the judgment of the researcher.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Study Success Case(Avoidance of ostomy) | 24 Weeks
  Study Success Case" is defined as a case which has met both the "Clinical Success" and "Technical Success" requirements throughout the 24 weeks (6 Months) monitoring period, following the initial surgical treatment with COLO-BT™ or temporary ileostomy

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Falvo, MD, Principal Investigator — Jacobs School of Medicine & Biomedical Sciences, State University of New York at Buffalo
Locations (3):
- United States (3):
  - Jacobs School of Medicine & Biomedical Sciences, State University of New York at Buffalo, Buffalo, New York
  - PennState Health - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Baylor College of Medicine, Houston, Texas